CLINICAL TRIAL: NCT02214459
Title: Dietary Approaches to Stopping Hypertension (DASH) Mobile App Pilot
Acronym: DASH Mobile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-32775
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
Keywords: mHealth; Hypertension; Mobile; smartphone; diet; lifestyle; bluetooth; physical acitvity; behavior change; motivational interviewing
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mhealth counseling (Experimental): DASH Mobile mhealth enhanced coaching
  Interventions: Behavioral: DASH Mobile mhealth enhanced coaching

INTERVENTIONS:
Behavioral: DASH Mobile mhealth enhanced coaching — Phone calls with a health coach that utilize the tracking data collected by the app and devices.

SUMMARY:
The enormous burden of hypertension (HTN) creates a need for effective, scalable, low risk interventions. The DASH program of diet and exercise based lifestyle change is the most well-established, evidence-based behavioral intervention to control HTN. Its recommendations are central to HTN control national guidelines and consumer health products aimed at behavioral management of HTN. However, translating these recommendations into population-wide, inexpensive, sustainable programs have to date proven largely unrealized. The objective of the proposed study is to determine the efficacy of a HTN intervention behavior change platform, 'DASH Mobile', in which patients with HTN receive counseling about the DASH diet, physical activity and HTN related behaviors from health coaches trained in evidenced-based behavioral counseling methods. DASH mobile has two primary components: 1) a smartphone app that captures patients' behavioral data using intuitive self-tracking for DASH diet intake and Bluetooth wireless sensors for blood pressure, weight and physical activity and 2) a web-based coaching portal through which health coaches view and respond to patients' behavioral data and assist them in setting goals for changing behaviors consistent with their HTN behavior change plan. We aim to conduct a pilot trial of 30 HTN patients to determine improvement from baseline to 3-month follow-up in physiological (blood pressure, weight); behavioral (diet & physical activity); and psychological (e.g., quality of life) measures over a 3-month intervention. Completing this research will result in preliminary feasibility and efficacy data for a larger randomized efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* hypertension
* prehypertension
* smartphone
* english speaking

Exclusion Criteria:

* on more than 1 medicine for hypertension
* live outside Boston metro area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States